CLINICAL TRIAL: NCT02793700
Title: Pharmacokinetics and Modeling of Betamethasone Therapy in Threatened Preterm Birth
Brief Title: Pharmacokinetics (PK) and Modeling of Betamethasone Therapy in Threatened Preterm Birth
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, David Haas, Dr, MD, MS, Indiana University
Other Study IDs: 1604640151
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Premature Labor
Keywords: Betamethasone
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal whole blood Cord blood Placenta
Oversight: Data Monitoring Committee: No

SUMMARY:
Respiratory distress syndrome (RDS) is a life-threatening condition for premature neonates. Antenatal glucocorticoids have been used clinically in women with threatened preterm birth to accelerate lung maturation for more than 40 years. The current treatment strategy for women with threatened preterm delivery is for a standard, "one size fits all" dosing with either betamethasone (BMZ) or dexamethasone. It is well known that pregnancy introduces additional variability in response to medication therapy with different physiological changes and alterations in the activity of drug metabolizing enzymes. The objective of this project is to evaluate the pharmacokinetic (PK), pharmacodynamic, and pharmacogenetic parameters of betamethasone (BMZ) and determine the differences in response and benefit in pregnancy. An individualized dosing approach to medications in pregnancy, such as BMZ, is crucial to optimize efficacy of this important medication.

DETAILED DESCRIPTION:
After consent, a maternal sample of whole blood will be obtained for DNA isolation. Investigators will collect plasma samples at 4 time points on all participants. These will be done at baseline (pre-dose), and 0.5-2 hours, 4-6 hours, and 22-24 hours after the first dose of BMZ is administered. Investigators will obtain serum for estriol measurement on all participants before or within 2 hours of antenatal corticosteroid administration and about 24 hours after each dose is given (betamethasone is administered as 2 doses 24 hours apart). Investigators will obtain a saliva sample for measurement of estriol at the same times. Participants will be offered optional participation in a more detailed PK portion of the study. Participants who consent to this part of the study will have additional plasma samples obtained at a schedule of sampling of approximately 10-15 hours after the first dose and then 6-8 hours, 24, and 48 hours after the 2nd dose. One sample will be collected at each of these times. At the time of delivery, umbilical cord blood will be collected before being discarded for DNA, serum and plasma. Four placenta sections will be collected. A maternal blood sample will also be obtained for serum and plasma. If the investigators are unable to obtain umbilical cord blood, a buccal swab will be collected from the baby for DNA extraction. A chart review will be done on the infant within 30 days of birth to review and record neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 23-34 weeks with a diagnosis of threatened preterm labor or preterm premature rupture of membranes, or other diagnosis with a high likelihood of preterm delivery where the provider is recommending administering antenatal corticosteroids
* Singleton gestation
* Live fetus at the time of enrollment
* Being administered antenatal corticosteroids to enhance lung maturity
* Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* Maternal age <18 years old
* Major congenital anomalies
* Known severe abruptio placentae at the time of enrollment
* Multiple gestations
* Hepatic failure (history of hepatic failure, cirrhosis or 2- fold increase in Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT)
* Renal failure (serum creatinine > 2 mg/dl)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women 18 years of age or older who are between 23-34 weeks gestation and being administered BMZ for fetal lung maturity.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2016-07; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Diagnosis of respiratory distress syndrome | up to 30 days of life
  The diagnosis of RDS made by the neonatologist staff based on clinical criteria

CONTACTS AND LOCATIONS:
Overall Officials: David M Haas, MD, MS, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Eskenazi Hospital, Indianapolis, Indiana
  - IUH Methodist Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Undecided
No plan for availability of individual participant data